CLINICAL TRIAL: NCT01878409
Title: Study of Sexuality in Parkinson Disease
Acronym: Sex-PD
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 652
Record Dates: First submitted 2013-06-06; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson Disease
Keywords: Sexuality; Parkinson Disease; BISF; IIEF; FSFI
MeSH Terms: conditions — Parkinson Disease; Sexuality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parkinson Disease: Patients with Parkinson Disease
- Healthy Subjects: Healthy Subjects

SUMMARY:
The aim of this study is to evaluate the different aspects of sexual function among adults with Parkinson Disease to develop a treatment and address sexual problems as a routine part of diagnostic workup and therapeutic planning.

DETAILED DESCRIPTION:
Because there is limited literature on sexual function in Parkinson disease, in this study, we examined sexual functioning in a large groups of patients with idiopathic Parkinson Disease compared with healthy subjects in the Italian community. To assess sexual function in PD we used the Brief Index of Sexual Functioning [(BISF-M for man; BISF-W for woman), the International Index of Erectile Function (IIEF) and the Female Sexual Function Index (FSFI). Participants were also assessed by the Beck Depression Inventory (BDI).

This study aimed to provide a thorough epidemiological description of sexual dysfunction in Parkinson's disease. The knowledge of sexual function in PD might help to plan effective interventionist measures and ultimately to optimize patient's and the partner's quality of life.

Parkinson patients (aged 40-80) and 123 healthy controls (aged 40-80) will be recruited from four Italian Movement Disorders Clinics.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD
* marital status
* age 40-80

Exclusion Criteria:

* patients taking PDE

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as having idiopathic PD were recruited from four Italian Movement Disorders Clinics
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
BISF | Baseline
  Brief Index of Sexual Functioning (BISF-M for man; BISF-W for woman)International Index of Erectile Function (IIEF) Female Sexual Function Index (FSFI)

SECONDARY OUTCOMES:
BDI | Baseline
  Beck Depression Inventory (BDI) is a 21.-item self report inventory, for measuring the severity of depression in clinical and nonclinical populations.
PDQ8 | Baseline
  Parkinson' Disease Questionnaire-8 (PDQ- 8) is a self completion PRO designed to address aspects of functioning and well-being for those affected by Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Priori, MD,PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Università di Milano
Locations (1):
- Fondazione IRCCS Ca' Granda, Milan, Italy, Italy